CLINICAL TRIAL: NCT02847117
Title: A Bioavailability Study of the Natural Chios Mastiha in Blood and Urine Samples of Healthy Adults.
Brief Title: Bioavailability of the Microconstituents of Natural Chios Mastiha in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, "Assistant Professor in Foods & Human Nutrition", Harokopio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Mastiha BIO-GR (304)
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Biological Availability
Keywords: Natural Mastiha, Bioavailability
MeSH Terms: interventions — mastiha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mastiha (Other)
  Interventions: Other: Mastiha

INTERVENTIONS:
Other: Mastiha — The volunteers will follow a low-phytochemical diet for five days, meaning that they will exclude fruits, vegetables, legumes, coffee, tea, alcoholic beverages and chocolate. On the day of the experiment and after overnight fasting, the volunteers will consume 10g of natural Mastiha and blood samples will be obtained on timepoints 0h, 30min, 1h, 2h, 4h, 6h and 24h after Mastiha intake. Until timepoint 6h, will be allowed to consume only water. Urine samples will also be collected on timepoints 0h, 4h, 8h and 24h.

SUMMARY:
Mastiha is a natural product from the tree Pistacia lentiscus var. Chia (Anacardiaceae) growing exclusively in the Southern part of Chios Island. It is the natural resinous exudate produced after longitudinal incisions made at close intervals from the base of the trunk up to the thicker branches of the tree. U.S. Food and Drug Administration has classified Mastiha as GRAS. Previous research demonstrates Mastiha's safety, as well as anti-inflammatory, antimicrobial and antioxidant properties. In addition, the European Medicine Agency has recently recognized Mastiha as a natural medicine and classified it to the category of traditional herbal medicines in diarrhea problems, mild dyspeptic disorders, skin inflammation and healing (EMA/HMPC/46758/2015).

However, the bioavailability of its microconstituents in human biological samples is still undetermined. To this end, the current study aims to investigate the whether Mastiha's compounds are bioavailable in healthy adults. Twenty apparently healthy men, aged 20-40 years old, will be enrolled based on certain inclusion and exclusion criteria. The staff of the study will provide detailed information regarding the aims, the methods, anticipated benefits and potential hazards of the study and all patients will receive the Patient Information Leaflet (PIL). Ample time (48 hours) will be provided in order to decide whether they want to participate in the protocol. Each patient agreeing to participate will sign an Informed Consent document and the staff will explain to patients that they are under no obligation to enter the trial and that they can withdraw at any time during the trial, without having to give a reason. A copy of the signed Informed Consent will be given to the participant.

After enrollment, the volunteers will undergo a medical and dietary assessment and their health status will be evaluated through a complete blood count. Then, they will follow a low-phytochemical diet for five days, meaning that they will exclude fruits, vegetables, legumes, coffee, tea, alcoholic beverages and chocolate. On the day of the experiment and after overnight fasting, the volunteers will consume 10g of natural Mastiha and blood samples will be obtained on timepoints 0h, 30min, 1h, 2h, 4h, 6h and 24h after Mastiha intake. Until timepoint 6h, they will be allowed to consume only water. Urine samples will also be collected on timepoints 0h, 4h, 8h and 24h.

After collection, the phenolic and terpenoid content or metabolites of Mastiha will be identified in plasma samples applying LC-HRMS. Additionally, the metabolomic profile will be assessed in plasma samples with LC-HRMS and in urine samples with NMR-based metabolomics. Oxidative stress will be evaluated through the CuSO4 technique and oxidised LDL levels in serum samples, as well as F-2 isoprostanes in urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40 years old
* BMI: 18.5-24.9 kg/m2

Exclusion Criteria:

* BMI > 25 kg/m2
* Alcohol or drug abuse
* Medication, vitamin or inorganic supplements
* Vegan or macrobiotic diet before and during the study
* Gastrointestinal diseases, such as IBD, peptic ulcer or GI cancer

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Phenolic and terpenoid content or metabolites of Mastiha identification | The phenolic and terpenoid content or metabolites of Mastiha will be identified in plasma samples applying LC-HRMS. Data will be presented through study completion, an average of 1 year.
Targeted and untargeted metabolic profile assessment | Plasma metabolites assessment with GC-MS, LC-HRMS and urine metabolites assessment with NMR will take place . Data will be presented through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Oxidative stress assessment | Serum resistance to oxidation will be assessed through the CuSO4 technique, oxidised LDL levels and uric acid levels. F-2 isoprostanes determination will take place in urine samples. Data will be presented through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Harokopio University, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romani A, Pinelli P, Galardi C, Mulinacci N, Tattini M. Identification and quantification of galloyl derivatives, flavonoid glycosides and anthocyanins in leaves of Pistacia lentiscus L. Phytochem Anal. 2002 Mar-Apr;13(2):79-86. doi: 10.1002/pca.627. PMID 12018027
- [Background] Kaliora AC, Dedoussis GV, Schmidt H. Dietary antioxidants in preventing atherogenesis. Atherosclerosis. 2006 Jul;187(1):1-17. doi: 10.1016/j.atherosclerosis.2005.11.001. Epub 2005 Nov 28. PMID 16313912
- [Background] Crowell PL. Prevention and therapy of cancer by dietary monoterpenes. J Nutr. 1999 Mar;129(3):775S-778S. doi: 10.1093/jn/129.3.775S. PMID 10082788
- [Background] Gonzalez-Burgos E, Gomez-Serranillos MP. Terpene compounds in nature: a review of their potential antioxidant activity. Curr Med Chem. 2012;19(31):5319-41. doi: 10.2174/092986712803833335. PMID 22963623
- [Background] Inouye S, Takizawa T, Yamaguchi H. Antibacterial activity of essential oils and their major constituents against respiratory tract pathogens by gaseous contact. J Antimicrob Chemother. 2001 May;47(5):565-73. doi: 10.1093/jac/47.5.565. PMID 11328766
- [Background] Inouye S, Yamaguchi H, Takizawa T. Screening of the antibacterial effects of a variety of essential oils on respiratory tract pathogens, using a modified dilution assay method. J Infect Chemother. 2001 Dec;7(4):251-4. doi: 10.1007/s101560170022. PMID 11810593
- [Background] Ohno T, Kita M, Yamaoka Y, Imamura S, Yamamoto T, Mitsufuji S, Kodama T, Kashima K, Imanishi J. Antimicrobial activity of essential oils against Helicobacter pylori. Helicobacter. 2003 Jun;8(3):207-15. doi: 10.1046/j.1523-5378.2003.00146.x. PMID 12752733
- [Background] Ding Y, Nguyen HT, Kim SI, Kim HW, Kim YH. The regulation of inflammatory cytokine secretion in macrophage cell line by the chemical constituents of Rhus sylvestris. Bioorg Med Chem Lett. 2009 Jul 1;19(13):3607-10. doi: 10.1016/j.bmcl.2009.04.129. Epub 2009 May 3. PMID 19447618
- [Background] Rodrigues TG, Fernandes A Jr, Sousa JP, Bastos JK, Sforcin JM. In vitro and in vivo effects of clove on pro-inflammatory cytokines production by macrophages. Nat Prod Res. 2009;23(4):319-26. doi: 10.1080/14786410802242679. PMID 19296372
- [Background] Andrikopoulos NK, Kaliora AC, Assimopoulou AN, Papapeorgiou VP. Biological activity of some naturally occurring resins, gums and pigments against in vitro LDL oxidation. Phytother Res. 2003 May;17(5):501-7. doi: 10.1002/ptr.1185. PMID 12748987
- [Background] Gioxari A, Kaliora AC, Papalois A, Agrogiannis G, Triantafillidis JK, Andrikopoulos NK. Pistacia lentiscus resin regulates intestinal damage and inflammation in trinitrobenzene sulfonic acid-induced colitis. J Med Food. 2011 Nov;14(11):1403-11. doi: 10.1089/jmf.2010.0240. Epub 2011 May 25. PMID 21612460
- [Background] Papalois A, Gioxari A, Kaliora AC, Lymperopoulou A, Agrogiannis G, Papada E, Andrikopoulos NK. Chios mastic fractions in experimental colitis: implication of the nuclear factor kappaB pathway in cultured HT29 cells. J Med Food. 2012 Nov;15(11):974-83. doi: 10.1089/jmf.2012.0018. Epub 2012 Aug 14. PMID 22891614
- [Background] Williamson G, Manach C. Bioavailability and bioefficacy of polyphenols in humans. II. Review of 93 intervention studies. Am J Clin Nutr. 2005 Jan;81(1 Suppl):243S-255S. doi: 10.1093/ajcn/81.1.243S. PMID 15640487
- [Background] Kountouri AM, Mylona A, Kaliora AC, Andrikopoulos NK. Bioavailability of the phenolic compounds of the fruits (drupes) of Olea europaea (olives): impact on plasma antioxidant status in humans. Phytomedicine. 2007 Oct;14(10):659-67. doi: 10.1016/j.phymed.2007.06.001. Epub 2007 Sep 17. PMID 17870451
- [Background] Kanellos PT, Kaliora AC, Liaskos C, Tentolouris NK, Perrea D, Karathanos VT. A study of glycemic response to Corinthian raisins in healthy subjects and in type 2 diabetes mellitus patients. Plant Foods Hum Nutr. 2013 Jun;68(2):145-8. doi: 10.1007/s11130-013-0348-y. PMID 23564595
- [Background] Lemonakis N, Magiatis P, Kostomitsopoulos N, Skaltsounis AL, Tamvakopoulos C. Oral administration of chios mastic gum or extracts in mice: quantification of triterpenic acids by liquid chromatography-tandem mass spectrometry. Planta Med. 2011 Nov;77(17):1916-23. doi: 10.1055/s-0031-1279996. Epub 2011 Aug 25. PMID 21870323